CLINICAL TRIAL: NCT03786198
Title: A 24 Weeks Activity Program in Patients With Early Breast Cancer Receiving Aromatase Inhibitor Therapy. A Multicenter Randomized Phase III Trial
Brief Title: Activity Program During Aromatase Inhibitor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAKK 95/17
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Early Breast Cancer
Keywords: early breast cancer; aromatase inhibitor therapy; activity program; physical activity; activity tracker; pedometer; stepcounter
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Commission on Professional and Hospital Activities

STUDY DESIGN:
Intervention Model Description: 1. Home-based walking intervention for 24 weeks + standard adjuvant AI therapy
  2. Physical activity according to standard recommendations for 24 weeks + standard adjuvant AI therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a) Home-based walking intervention (Experimental): Home-based walking intervention, wearing a wrist worn activity tracker, for 24 weeks + standard adjuvant AI therapy
  Interventions: Behavioral: Activity program
- b) Physical activity according to standard recommendations (Active Comparator): Physical activity according to standard recommendations, wearing a wrist worn activity tracker (with no feedback about performed activity), for 24 weeks + standard adjuvant AI therapy
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Activity program — Home-based walking intervention, wearing a wrist worn activity tracker, for 24 weeks
  Arms: a) Home-based walking intervention
Behavioral: Control — Physical activity according to standard recommendations, wearing a wrist worn activity tracker (with no feedback about performed activity), for 24 weeks + standard adjuvant AI therapy
  Arms: b) Physical activity according to standard recommendations

SUMMARY:
The primary aim of the trial is to investigate if a simple outdoor walking intervention, which is practicable under real-life conditions, beginning at the start of adjuvant aromatase inhibitor (AI) therapy, can prevent the occurrence of muscle or joint pain/stiffness in breast cancer patients.

DETAILED DESCRIPTION:
After tumor removal, patients with hormone receptor positive breast cancer tumors often receive adjuvant endocrine treatment, with the use of an aromatase inhibitor (AI) being standard of care in the population of postmenopausal women. Common side effects of AI therapy are joint pain, muscle pain, stiffness, fatigue, hot flashes, and weight gain. Arthralgia and/or myalgia can result in lower physical activity and can negatively influence quality of life (QoL). In addition, muscle or joint pain/stiffness are among the main reasons for non-compliance and discontinuation of AI therapy. Because AI therapy is usually administered for 5 and sometimes even 10 years, this is a major clinical challenge.

For breast cancer patients undergoing AI therapy, physical activity can provide potential benefit by reducing muscle/joint pain and fatigue and can thus improve QoL. The preventive effect of physical activity on AI side effects, however, remains elusive. In addition, activity programs to reduce AI side effects have so far mostly been rather complex. The primary aim of the trial is to investigate if a simple outdoor walking intervention, which is practicable under real-life conditions, beginning at the start of adjuvant AI therapy, can prevent the occurrence of muscle or joint pain/stiffness in breast cancer patients.

Furthermore, this trial will assess the effect of physical activity on symptom burden in general and quality of life in patients receiving adjuvant AI therapy. During the follow-up phase, the trial will assess whether this intervention leads to a sustained change in lifestyle regarding activity, less pain, and better treatment adherence in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures.
* Histologically confirmed hormone-receptor-positive newly diagnosed breast cancer, AJCC (American Joint Committee on Cancer) stage I-III
* Patient had tumor removal by breast conserving surgery or mastectomy, followed by chemotherapy (if indicated) and/or radiotherapy (if indicated)
* Patient is starting adjuvant first-line endocrine treatment with an AI alone (in postmenopausal women) or combined endocrine treatment with an AI and ovarian suppression with an LHRH-agonist (in premenopausal women)
* Patient completed the PRO Form Eligibility before registration
* Patient is fluent in German, Italian, or French
* Patient is willing to wear a wrist worn activity tracker for 24 weeks
* Female patient, age ≥ 18 years
* WHO performance status 0-2

Exclusion Criteria:

* Pre-existing severe medical conditions such as heart or lung problems or musculoskeletal conditions precluding participation in the physical activity program of moderate walking a total of 150 minutes per week as determined by the local investigator
* Mild, moderate, or severe pain (other than post-operative pain) in the last 24 hours due to muscle/joint pain on the BPI-SF single item "worst pain" ("worst pain" ≥3) within 7 days prior to registration
* Inoperable, locally advanced and/or metastatic breast cancer
* Active rheumatoid arthritis
* Neoadjuvant endocrine treatment with an AI
* NSAIDs, acetaminophen or opioids on a regular basis (> 1 time per week)
* Concurrent participation in other clinical trials or observational studies
* Any other serious psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the intervention and follow-up or affect patient compliance with trial procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Incidence of muscle or joint pain/stiffness as measured by BPI-SF single-item worst pain score | Up to 24 weeks after randomization
  Muscle or joint pain/stiffness will be assessed at baseline, 3, 9, 12, 15, 18, 21, 24 weeks after randomization by the BPI-SF questionnaire.
  The BPI-SF is a 14-item self-administered questionnaire which is routinely used in clinical trials to assess pain severity and pain interference with daily activities in patients with cancer. Pain severity is assessed by four items including pain at its "worst", "least", "average" in the last 24 hours and "now" (current pain), each item being rated on a 0-10 scale.

SECONDARY OUTCOMES:
Fatigue | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Fatigue will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
QoL: Physical scale (EORTC QLQ-C30) | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Physical scale will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
QoL: Rose scale (EORTC QLQ-C30) | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Role scale will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
QoL: Emotional scale (EORTC QLQ-C30) | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Emotional scale will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
QoL: Cognitive scale (EORTC QLQ-C30) | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Cognitive scale will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
QoL: Social functioning scale (EORTC QLQ-C30) | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Cognitive scale will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Nausea/Vomiting | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Nausea/vomiting will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Pain (EORTC QLQ-C30) | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Pain will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Global health status | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Global health status will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Dyspnoea | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Dyspnoea will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Insomnia | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Insomnia will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Appetite loss | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Appetite loss will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Constipation | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Constipation will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Diarrhoea | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Diarrhoea will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Financial difficulties | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Financial difficulties will be assessed at baseline, during intervention phase and during follow-up phase using the corresponding symptom scale of the EORTC QLQ-C30 version 3.0.
Hot flashes | Baseline, 12 and 24 weeks and 1 and 2 years after randomization
  Hot flashes will be assessed at baseline, during intervention phase and during follow-up phase via the item 37 of the EORTC QLQ BR-23.
Intensity of muscle or joint pain/stiffness and its impact on everyday functioning | Baseline, 3, 9, 12, 15, 18, 21, 24 weeks and 1, 2 years after randomization
  Severity of muscle or joint pain/stiffness will be measured by the four BPI pain severity items. Pain interference will be calculated as the mean of the seven interference items.
Walking activity | Baseline, 3, 9, 12, 15, 18, 21, 24 weeks after randomization
  During trial intervention phase, daily steps will be measured by a wrist worn activity tracker.
AI treatment adherence (diary) | Baseline, 3, 9, 12, 15, 18, 21, 24 weeks.
  Adherence will be assessed by patient self-report (diary).
AI treatment adherence (questionnaire) | Baseline, 12, 24 weeks and 1, 2 years after randomization
  Adherence will be assessed by patient self-report (questionnaire completed at visits).

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Honecker, MD, Study Chair — Tumor- und Brustzentrum ZeTuP St.Gallen; Nicolette Hoefnagels, MSc, Study Chair — Tumor- und Brustzentrum ZeTuP St.Gallen
Locations (32):
- Switzerland (32):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - CABA - Zentrum für Onkologie, Psychologie und Bewegung, Basel
  - Brustzentrum Basel - Praxis für ambulante Tumortherapie, Basel
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Hirslanden Brustzentrum Bern Biel, Bern
  - Clinique des Grangettes, Centre du sein, Chêne-Bougeries
  - Kantonsspital Graubünden, Chur
  - Tumorzentrum ZeTuP Chur, Chur
  - Brustzentrum Thurgau, Frauenfeld
  - Centre du sein Fribourg / Brustzentrum Freiburg, Fribourg
  - Clinique De Genolier, Genolier
  - FOLM - Fondazione Oncologia Lago Maggiore, Locarno
  - Hirslanden Klinik St. Anna, Lucerne
  - Oncologia Varini&Calderoni&Christinat, Lugano
  - Kantonsspital Luzern, Luzerne
  - Onkologie Zentrum Spital Männedorf, Manno
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Mendrisio
  - Hôpital Neuchâtelois, Neuenhof
  - Kantonsspital Olten, Olten
  - Tumorzentrum ZeTuP Rapperswil-Jona, Rapperswil-Jona
  - Tumorzentrum ZeTUP, Sankt Gallen
  - Brustzentrum Ostschweiz, Sankt Gallen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Rundum Onkologie am Bahnhofpark, Sargans
  - Hôpital de Sion, Sion
  - Regionalspital Thun, Thun
  - Kantonsspital Winterthur, Brustzentrum, Winterthur
  - Onkologie Bellevue, Zurich
  - Brustzentrum Zürich, Zurich
  - Universitäts Spital Zürich, Zurich